CLINICAL TRIAL: NCT05013840
Title: Opinions of Healthcare Providers About Neuromodulation for Pain: an Online Survey
Brief Title: Opinions of Healthcare Providers About Neuromodulation
Status: Completed | Type: Observational
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: INCEPTION
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Neuromodulation; Pain; Survey
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians using neuromodulation
  Interventions: Behavioral: Filling in an online survey

INTERVENTIONS:
Behavioral: Filling in an online survey — Physicians are asked to fill in an online survey regarding 1) goals to treat patients with neuromodulation for pain, 2) factors that respondents expect to change according to neuromodulation for pain and 3) their definition of success of neuromodulation for pain.

SUMMARY:
The goal of this online survey is to gain further insight in the goals, expectations and definition of success for neuromodulation for pain, according to healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

- Male and female adults who are involved in the management of chronic pain and more specifically in neuromodulation for pain (including but not limited to anesthesiologists, neurosurgeons, nurses).

Exclusion Criteria:

- Not involved in management of chronic pain through neuromodulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female adults who are involved in the management of chronic pain and more specifically in neuromodulation for pain (including but not limited to anesthesiologists, neurosurgeons, nurses).The survey will be spread at the 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris from 2/9/2021 to 4/9/2021.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Physician goals, evaluated with a self-constructed question. | Cross-sectional evaluation during 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris in September.
  Goals of physicians to treat patients with neuromodulation for pain.
Physician expectations, evaluated with a self-constructed question. | Cross-sectional evaluation during 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris in September.
  Factors that respondents expect to change according to neuromodulation for pain.
Physician definition of success, evaluated with a self-constructed question. | Cross-sectional evaluation during 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris in September.
  Physician definition of success of neuromodulation for pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

REFERENCES:
- [Derived] Goudman L, De Smedt A, Billot M, Roulaud M, Rigoard P, Moens M. Opinions of Health Care Providers About Neuromodulation for Pain: Results of an Online Survey at the 2nd Joint Congress of the International Neuromodulation Society European Chapters. Neuromodulation. 2023 Dec;26(8):1887-1892. doi: 10.1016/j.neurom.2022.04.038. Epub 2022 May 10. PMID 35551866